CLINICAL TRIAL: NCT01235520
Title: Phase III, Multi-center, Randomized, 12-week, Double-blind, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of RO4917838 in Patients With Sub-optimally Controlled Symptoms of Schizophrenia Treated With Antipsychotics Followed by a 40-week Double-blind, Parallel-group, Placebo-controlled Treatment Period.
Brief Title: A Study of RO4917838 in Patients With Sub-optimally Controlled Symptoms of Schizophrenia (NN25307)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN25307; 2010-020696-23
Record Dates: First submitted 2010-10-22; First posted 2010-11-05 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-06

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: RO4917838
- 2 (Experimental)
  Interventions: Drug: RO4917838
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Oral doses, once a day for 52 weeks
  Arms: 3
Drug: RO4917838 — Oral dose level 1, once a day for 52 weeks
  Arms: 1
Drug: RO4917838 — Oral dose level 2, once a day for 52 weeks
  Arms: 2

SUMMARY:
This randomized, multi-center, double-blind, parallel-group, placebo-controlled study will evaluate the efficacy and safety of RO4917838 in patients with sub-optimally controlled symptoms of schizophrenia. Patients, on stable treatment with antipsychotics, will be randomized to receive daily oral doses of RO4917838 or matching placebo for 52 weeks, followed by an optional treatment extension for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Diagnosis of schizophrenia
* Clinical stability for 16 weeks (4 months) prior to randomization
* Antipsychotic treatment stability for the past 12 weeks prior to randomization
* With the exception of clozapine, patients are on any of the available marketed atypical or typical antipsychotic (treatment with a maximum of two antipsychotics)

Exclusion Criteria:

* Has treatment resistant schizophrenia as judged by the treating physician OR have failed two trials
* Evidence that patient has clinically significant uncontrolled or unstable medical disorder (e.g. cardiovascular, renal hepatic, gastrointestinal, hematologic, immunological, neurological, endocrine, metabolic or pulmonary disease)
* Patient has a body mass index (BMI) of <17 or >40 kg/m2, respectively
* Diagnosis of mental retardation or severe organic brain syndromes
* In the investigator's judgment, a significant risk of suicide or violent behavior

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2011-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Positive symptoms factor score assessed by Positive and Negative Syndrome Scale (PANSS) | Change from baseline to Week 12
Safety (incidence of adverse events) | Week 12

SECONDARY OUTCOMES:
Symptom domains of schizophrenia using Positive and Negative Syndrome Scale (PANSS) | Change from baseline to Week 12
Disease improvement on Clinical Global Impression - Improvement (CGI-I) symptoms scale | Change from baseline to Week 12
Disease severity on Clinical Global Impression - Severity (CGI-S) symptoms scale | Change from baseline to Week 12
Safety (incidence of adverse events) | 60 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (93):
- United States (27):
  - Little Rock, Arkansas
  - Buena Park, California
  - Cerritos, California
  - Downey, California
  - La Palma, California
  - Pasadena, California
  - Pico Rivera, California
  - Miami, Florida
  - Marietta, Georgia
  - Oak Brook, Illinois
  - Iowa City, Iowa
  - Glen Burnie, Maryland
  - Las Vegas, Nevada
  - Toms River, New Jersey
  - Willingboro, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Fresh Meadows, New York
  - New York, New York
  - Raleigh, North Carolina
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Scranton, Pennsylvania
  - Bellaire, Texas
  - Dallas, Texas
  - The Woodlands, Texas
  - Kirkland, Washington
- Argentina (7):
  - Buenos Aires
  - Ciudad Autonoma Bs As
  - Córdoba
  - La Plata
  - Mendoza
  - Rosario
  - Santiago del Estero
- Australia (4):
  - Westmead, New South Wales
  - Clayton, Victoria
  - Frankston, Victoria
  - Melbourne, Victoria
- Colombia (3):
  - Barranquilla
  - Bello
  - Bogotá
- Finland (2):
  - Helsinki
  - Kuopio
- France (6):
  - Clermont-Ferrand
  - Dole
  - Élancourt
  - Marseille
  - Strasbourg
  - Toulon
- Hungary (4):
  - Balassagyarmat
  - Budapest
  - Győr
  - Gyula
- India (8):
  - Ahmedabad
  - Bangalore
  - Jaipur
  - Kalyān
  - Mangalore
  - Nashik
  - Pune
  - Vadodara
- Mexico (3):
  - México
  - Monterrey
  - San Luis Potosí City
- Romania (7):
  - Arad
  - Bucharest
  - Cluj-Napoca
  - Lasi
  - Oradea
  - Sibiu
  - Targouiste
- Russia (10):
  - Kemerovo
  - Lipetsk
  - Moscow
  - Moscow Region
  - Nizhny Novgorod
  - Saint Petersburg
  - Samara
  - Sartatov
  - Talagi
  - Tomsk
- South Korea (6):
  - Busan
  - Gwangju
  - Gyeonggi-do
  - Incheon
  - Jeollabuk-do
  - Seoul
- Sweden (3):
  - Malmo
  - Stockholm
  - Uppsala
- United Kingdom (3):
  - Edinburgh
  - London
  - Oxford

REFERENCES:
- [Derived] Bugarski-Kirola D, Iwata N, Sameljak S, Reid C, Blaettler T, Millar L, Marques TR, Garibaldi G, Kapur S. Efficacy and safety of adjunctive bitopertin versus placebo in patients with suboptimally controlled symptoms of schizophrenia treated with antipsychotics: results from three phase 3, randomised, double-blind, parallel-group, placebo-controlled, multicentre studies in the SearchLyte clinical trial programme. Lancet Psychiatry. 2016 Dec;3(12):1115-1128. doi: 10.1016/S2215-0366(16)30344-3. Epub 2016 Nov 2. PMID 27816567